CLINICAL TRIAL: NCT00155623
Title: Establish the Precise Epidemiologic Data of Helicobacter Pylori Infection in Children and Adolescents - Using the 13C-Urea Breath Test
Brief Title: Establish Epidemiologic Data of H. Pylori Infection in Children and Adolescents-Using C13-UBT
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Other Study IDs: 24642; DOH90-DC-1031; DOH91-DC-1021; DOH92-DC-1051
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2001-01

CONDITIONS: H. Pylori Infection
Keywords: H. pylori, 13C-urea breath test, serology, epidemiology

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The aims of this prospective study are: (1) to prospectively investigate the "true" prevalence rate, the acquisition and spontaneous clearance of H. pylori infection year by year in the population whose ages between seven and fifteen. (2) to explore the risk factors of transmission of H. pylori infection in Taiwan. (This information may be use as the guide for conduction of the national policy of public health and disease prevention.)

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori), a spiral microaerophilic Gram-negative bacterium isolated in 1983, is now known as the most common gastrointestinal bacterial infection worldwide. It is the principal cause of chronic gastritis and is strongly associated with peptic ulcer disease as well as gastric cancer, including gastric lymphoma (MALT type). In developed countries, infection occurs in more than 50% of adults, whereas developing countries have infection rates reaching 90%. Among those with H. pylori infection, eradication therapy alters the natural history of recurrences with attendant morbidity and death, which previously required lifelong maintenance therapy. Perhaps the greatest concern with regard to infection with H. pylori is the increased risk for the development of gastric cancers in adulthood. This is particularly relevant because infection dating from childhood appears to enhance the risk of carcinogenesis. Because H. pylori infection is contracted primarily during the childhood years, additional epidemiological studies among pediatric populations are imperative. Therefore the validation of an inexpensive, easy-to perform, sensitive, specific, and noninvasive diagnostic test for H. pylori infection in children and adolescents is of paramount importance to enhance our presently limited understanding of H. pylori-related diseases. The optimal noninvasive tests for epidemiological research of H. pylori infection in children are still not well identified. Serologic immunoassays based on H. pylori antigens require validation in the pediatric population under evaluation. As the result of our previous study, the serological test was not sensitive enough as an epidemiology screening tool for H. pylori infection in children.The aims of this prospective study are: (1) to prospectively investigate the "true" prevalence rate, the acquisition and spontaneous clearance of H. pylori infection year by year in the population whose ages between seven and fifteen. (2) to explore the risk factors of transmission of H. pylori infection in Taiwan. (This information may be use as the guide for conduction of the national policy of public health and disease prevention.) The study population will include students of one primary school and one junior high school in Lo-Tong area. There will be 150-160 cases in each age group and will be continuously followed-up for 3 years. Blood sample will be collected from each student for the serological test. 13C-urea breath test will be performed in each student, too. The parents of students will answer a questionnaire concerning the basic epidemiological data and possible factors related to the transmission of H. pylori. The students having new acquisition of H. pylori infection in the 2nd or 3rd years' follow-up period will be collected for further investigation. These student and their family will be invited to receive panendoscopy for the evaluation of possible pathology of stomach and the isolation H. pylori strain. These H. pylori isolates will be identified by molecular genotyping for the detection of possible source of transmission in the family. All of these results will be analyzed by a SAS system.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 15 years, both male and female. Teachers as adult control.

Exclusion Criteria:

* none

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000
Dates: Start 2001-02; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D., Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan